CLINICAL TRIAL: NCT03561597
Title: Pilot Evaluation of a Mobile Health Intervention to Identify Early Responders to Treatment in Adolescent Obesity as a Triage Approach
Brief Title: Mobile Health Intervention to Identify Early Responders to Treatment in Adolescent Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: National Institute of Education, Singapore (Other); National Dental Centre, Singapore (Other); Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 006100317
Record Dates: First submitted 2018-03-07; First posted 2018-06-19 (Actual); Results first posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2018-04

CONDITIONS: Adolescent Obesity
Keywords: stepped care; mobile application
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: prospective single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile health application (Experimental): Participants will undergo Kurbo program, a Mobile health application, for more detailed dietary and physical activity recommendations and implementation of behavioural changes. The patient's progress will be reviewed by the nurse clinician at one month post intervention to determine whether the BMI percentile has shown a reduction through the Kurbo Program. Patients that declined Kurbo intervention, has a BMI of more than 99th percentile or continue to have increase in their BMI percentile in Kurbo program, will be offered the high risk weight management clinic appointment for a more detailed multidisciplinary evaluation for targeted intervention. Patients that are able to engage with Kurbo intervention and showed a decrease in BMI percentile over 4 sessions of Kurbo will be offered the low risk weight management clinic (WMC). There will be a month 3 and month 6 visit for study measurements in this study.
  Interventions: Behavioral: Mobile health intervention

INTERVENTIONS:
Behavioral: Mobile health intervention — The Kurbo program is a multifunctional mobile application that aid adolescents and their families to learn healthy eating habits and weight management through the use of a mobile application with dietary self-monitoring and weekly interactive coaching sessions. Using the Kurbo app, adolescents track their food and exercise, as well as learn about healthy behaviours through games and videos. The Kurbo coaches check in with adolescents for 15 minutes once a week via video, phone or text over a 12 weeks period.

SUMMARY:
Background: The Expert Committee on the Assessment, Prevention and Treatment of Child and Adolescent Overweight and Obesity recommends a staged based approach to the management of adolescents with overweight and obesity from Stage 1-4 with increasing intensity of management in higher stages. Mobile health application is an attractive community based treatment for adolescent obesity due to its wide penetration and convenience. Early weight loss has been found to be the strongest predictor of good long term outcome in obesity. However there is currently no known study that use early weight loss as a predictor factor for a stepped up approach using a mobile health application.

Clinical significance: The current study use a mobile health intervention to identify participants with early weight loss in a stepped up approach.

Primary objective will be to examine the proportion of patients triaged to the low risk Weight Management Clinics (WMC) after brief intervention by a nurse coordination and completion of 4 sessions of Kurbo Program over a 12 month recruitment period.

Secondary objectives will be to examine changes in BMI z-score, metabolic profile, examine program feasibility and fidelity and explore other predictors of poor response to program.

Methodology:

Children aged 13-17 years old with BMI percentile of above 90th percentile, who are referred to the WMC, will receive a brief intervention by the WMC nurse coordinator followed by introduction to Kurbo program, a multifunctional mobile application, for more detailed dietary and physical activity recommendations and implementation of behavioural changes. Patients that are able to engage with Kurbo intervention and showed a decrease in BMI percentile over 4 sessions of Kurbo will be offered the low risk weight management clinic.

At baseline, month 3 and month 6, the patient's weight and height, body fat composition, waist circumference and blood pressure will be measured as per usual standard protocol. Questionnaires to assess eating, quality of life and dietary recall will be administered as part of the research. Accelerometers will also be fitted to assess physical activity.

At baseline and month 6, metabolic blood tests (HbA1C, fasting lipid panel, oral glucose tolerance test, fasting insulin level and liver function test) were collected after a minimum 8 hour fasting period together with bloods for aromatic amino acid, branch chain amino acid and long chain acylcarnitines .

Current low risk WMC patients will be offered 2 monthly follow up with optional dietician and exercise physiologists counselling and exercise sessions. The high risk WMC patients will be routinely offered the standard high risk follow up protocol consisting of weekly follow up with the multidisciplinary team for 4 weeks followed by 2 weekly appointments for 2 months and monthly appointment thereafter based on clinical response.

ELIGIBILITY:
Inclusion Criteria:

1. Overweight as defined by BMI percentile of above 90th percentile
2. Age 13-17 years old in the year of referral
3. Ability to provide informed consent
4. Adolescents with a phone which is able to download the application to be used on their devices

Exclusion Criteria:

1. Patients with secondary causes of obesity especially genetic syndromes e.g. Trisomy 21, Prader-Willi
2. Currently participating in a weight management program
3. Unable to understand and speak English sufficiently to give informed consent and complete the research assessments.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Chew, MBBS, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KKWCH, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Not available to other researchers

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mobile Health Application
Started | 40 (Recruited)
3 Month Follow up | 21 (Attended 3 month follow up)
Completed | 20 (Attend month 6 follow up)
Not Completed | 20
Not completed — Lost to Follow-up | 20

BASELINE CHARACTERISTICS:
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.8 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0
  Race: Asian | 40
  Race: Native Hawaiian or Other Pacific Islander | 0
  Race: Black or African American | 0
  Race: White | 0
  Race: More than one race | 0
  Race: Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 18
  Malay | 13
  Indian | 5
  Other | 4
Region of Enrollment [Number; unit: participants]
  Singapore | 40
Body Mass Index z scores [Mean (Standard Deviation); unit: BMI z score] | 2.07 (0.30)
Body Mass [Mean (Standard Deviation); unit: kg] | 81.2 (17.2)
Height [Mean (Standard Deviation); unit: cm] | 161.9 (11.4)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 30.7 (3.9)
Waist-height ratio [Mean (Standard Deviation); unit: ratio] | 0.61 (0.055)
Body fat percentage [Mean (Standard Deviation); unit: percentage] | 43.3 (5.9)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 121 (13)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 69 (9)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Triaged to the Low Risk Weight Management Clinics
Description: Examine the proportion of patients triaged to the low risk weight management clinics after brief intervention by a nurse coordination and completion of 4 sessions of Kurbo Program.
Time Frame: 6 month
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 40
Participants | 28

2. Secondary Outcome: Kurbo Program Feasibility, Percentage of Participants Who Completed at Least One Health Coaching Session
Description: To examine the feasibility of using Kurbo program as a waitlist intervention for the target population as measured by quantifying the percentage of patients offered the program who agreed to enrol and engaged in Kurbo coaching session
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 40
Participants | 33

3. Secondary Outcome: Kurbo Program Fidelity
Description: To examine program fidelity as measured by the percentage of patients who complete all of the 12 sessions of online coaching by Kurbo coaches, as part of Kurbo programme.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 40
Participants | 7

4. Secondary Outcome: Attrition Rate
Description: To examine the rate of attrition from weight management clinic after implementation of the waitlist intervention and new model of care in weight management clinic.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 40
Participants | 20

5. Secondary Outcome: Change in Weight From Baseline to 6 Months
Description: Change in weight from baseline to 6 months
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 20
kg | 3.59 [1.45 to 5.71]

6. Secondary Outcome: Change in Weight From Baseline to 3 Months
Description: Change in weight from baseline to 3 months
Time Frame: Baseline and 3 months
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 21
kg | 2.7 [0.5 to 4.8]

7. Secondary Outcome: Changes in Treatment Outcomes Using BMI Z-score
Description: To examine changes in treatment outcomes as a function of program fidelity as measured by those who complete more online coaching show greater improvements in BMI z-score. Body mass index (BMI) will be calculated as kg/m2 and BMI-z score calculated using the L, M, S parameters published by the Centre for Disease Control and Prevention. BMI z-score are measures of relative weight adjusted for child age and sex. Reduction of more than 0.25 in childhood obesity has been found to be clinically significant for reduction of cardiovascular risk factors.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: BMI z score
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 20
BMI z score | 0.035 [-0.028 to 0.098]

8. Secondary Outcome: Changes in Treatment Outcomes Using BMI Z-score From Baseline to 3 Months
Description: as for outcome 7
Time Frame: Baseline and 3 months
Measure: Mean (95% Confidence Interval); unit: BMI z-score
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 21
BMI z-score | 0.045 [-0.024 to 0.114]

9. Secondary Outcome: Change in %BMIp95 From Baseline to 6 Months
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 20
percentage | 4.53 [0.63 to 8.42]

10. Secondary Outcome: Change in %BMIp95 From Baseline to 3 Months
Time Frame: Baseline and 3 months
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 21
percentage | 4.3 [-0.83 to 9.47]

11. Secondary Outcome: Change in Waist Circumference From Baseline to 6 Months
Description: Change in waist circumference from Baseline to 6 months
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 20
cm | 0.3 [-2.6 to 3.2]

12. Secondary Outcome: Change in Waist Circumference From Baseline to 3 Months
Description: Change in waist circumference from Baseline to 3 months
Time Frame: Baseline and 3 months
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 21
cm | 1.1 [-1.9 to 4.2]

13. Secondary Outcome: Change in Waist to Height Ratio From Baseline to 6 Months
Description: To examine the effect of the waitlist intervention and WMC intervention on waist to height ratio at baseline and 6 months. Waist and height will be measured in cm and ratio of more than 0.5 is indicative of higher cardiometabolic risk. Reduction of the waist height ratio has been shown to be beneficial in cardiometabolic outcomes.
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: waist-height ratio
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 20
waist-height ratio | 0.004 [-0.014 to 0.022]

14. Secondary Outcome: Change in Waist to Height Ratio From Baseline to 3 Months
Description: To examine the effect of the waitlist intervention and WMC intervention on waist to height ratio at baseline and 3 months. Waist and height will be measured in cm and ratio of more than 0.5 is indicative of higher cardiometabolic risk. Reduction of the waist height ratio has been shown to be beneficial in cardiometabolic outcomes.
Time Frame: Baseline and 3 months
Measure: Mean (95% Confidence Interval); unit: waist-height ratio
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 21
waist-height ratio | -0.003 [-0.20 to 0.015]

15. Secondary Outcome: Change in Body Fat Percentage From Baseline to 6 Months
Description: Change in body fat percentage from Baseline to 6 months. Body fat percentage was assessed using a bioimpedance analysis.
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 20
percentage | -2.0 [-3.6 to 0.38]

16. Secondary Outcome: Change in Body Fat Percentage From Baseline to 3 Months
Description: Change in body fat percentage from Baseline to 3 months. Body fat percentage was assessed using a bioimpedance analysis.
Time Frame: Baseline and 3 months
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 21
percentage | -1.31 [-2.47 to -0.15]

17. Secondary Outcome: Changes in Systolic Blood Pressure Measurements From Baseline to 6 Months
Description: Changes in systolic blood pressure at baseline and 6 month measured in mmHg
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 19
mmHg | -2.1 [-6.8 to 2.5]

18. Secondary Outcome: Changes in Systolic Blood Pressure Measurements From Baseline to 3 Months
Description: Changes in systolic blood pressure at baseline and 3 month measured in mmHg
Time Frame: Baseline and 3 months
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 21
mmHg | -5.5 [-9.8 to -1.2]

19. Secondary Outcome: Changes in Diastolic Blood Pressure Measurements From Baseline to 6 Months
Description: Changes in diastolic blood pressure at baseline and 6 month measured in mmHg
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 20
mmHg | -3.2 [-7.3 to 0.85]

20. Secondary Outcome: Changes in Diastolic Blood Pressure Measurements From Baseline to 3 Months
Description: Changes in diastolicblood pressure at baseline and 3 month measured in mmHg
Time Frame: Baseline and 3 months
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 21
mmHg | -4.2 [-8.1 to -0.2]

21. Secondary Outcome: Changes in Nutrition From Baseline to 6 Months
Description: To examine the effects of waitlist intervention on nutrition using a three day food diary at baseline and 6 months to assess total caloric intake and number of servings of fruits and vegetables.
Time Frame: Baseline and 6 months
Population: Total kcal intake
Measure: Mean (95% Confidence Interval); unit: kcal
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 20
kcal | -332 [-598 to -66]

22. Secondary Outcome: Changes in Nutrition From Baseline to 3 Months
Description: To examine the effects of waitlist intervention on nutrition using a three day food diary at baseline and 3 months to assess total caloric intake and number of servings of fruits and vegetables.
Time Frame: Baseline and 3 months
Measure: Mean (95% Confidence Interval); unit: kcal
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 21
kcal | -300 [-576 to -24]

23. Secondary Outcome: Changes in Servings of Vegetables From Baseline to 6 Months
Description: To examine the effects of waitlist intervention on nutrition using a three day food diary at baseline and 6 months to assess number of servings of vegetables per day.
Time Frame: Baseline and 6 Months
Measure: Mean (95% Confidence Interval); unit: servings
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 20
servings | -0.0 [-0.4 to 0.4]

24. Secondary Outcome: Changes in Servings of Vegetables From Baseline to 3 Months
Description: To examine the effects of waitlist intervention on nutrition using a three day food diary at baseline and 3 months to assess number of servings of vegetables per day.
Time Frame: Baseline and 3 Months
Measure: Mean (95% Confidence Interval); unit: servings
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 21
servings | -0.17 [-0.5 to 0.1]

25. Secondary Outcome: Changes in Physical Activity From Baseline to 6 Months
Description: To examine the effects of waitlist intervention on physical activity using results from accelerometer to assess time spent on sedentary and moderate to vigorous physical activity at baseline and 6 months. The Actigraph data were processed using the Actilife 6 software. The Puyau cut-off point of 3200 counts per minute (cpm) was used to estimate time spent in moderate-to-vigorous physical activity (MVPA).
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: minutes in MVPA
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 20
minutes in MVPA | 5.3 [0.88 to 9.75]

26. Secondary Outcome: Changes in Physical Activity From Baseline to 3 Months
Description: To examine the effects of waitlist intervention on physical activity using results from accelerometer to assess time spent on sedentary and moderate to vigorous physical activity at baseline and 3 months. The Actigraph data were processed using the Actilife 6 software. The Puyau cut-off point of 3200 counts per minute (cpm) was used to estimate time spent in moderate-to-vigorous physical activity (MVPA).
Time Frame: Baseline and 3 months
Measure: Mean (95% Confidence Interval); unit: minutes in MVPA
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 21
minutes in MVPA | 1.47 [-4.3 to 7.2]

27. Secondary Outcome: Changes in Total Quality of Life From Baseline to 6 Months
Description: To examine the effects of waitlist intervention on quality of life at baseline and 6 months using Pediatric Quality of Life Inventory (PedsQL; UK version 4) will be administered as a comprehensive and multi-dimensional construct that includes physical, emotional, and social functioning to assess quality of life in the adolescents. The self-report scale had a five-point response scale (0 = never a problem, 1 = almost never, 2 = sometimes, 3 = often and 4 = almost always). Items are linearly transformed to a 0-100 scale, so that higher scores indicate better quality of life.
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 20
score on a scale | 1.4 [-4.2 to 7.0]

28. Secondary Outcome: Changes in Total Quality of Life From Baseline to 3 Months
Description: To examine the effects of waitlist intervention on quality of life at baseline and 3 months using Pediatric Quality of Life Inventory (PedsQL; UK version 4) will be administered as a comprehensive and multi-dimensional construct that includes physical, emotional, and social functioning to assess quality of life in the adolescents. The self-report scale had a five-point response scale (0 = never a problem, 1 = almost never, 2 = sometimes, 3 = often and 4 = almost always). Items are linearly transformed to a 0-100 scale, so that higher scores indicate better quality of life.
Time Frame: Baseline and 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 21
units on a scale | 2.4 [-3.1 to 7.9]

29. Secondary Outcome: Changes in Physical Domain of Quality of Life From Baseline to 6 Months
Description: To examine the effects of waitlist intervention on quality of life, physical domain, at baseline and 6 months using Pediatric Quality of Life Inventory (PedsQL; UK version 4). The self-report scale had a five-point response scale (0 = never a problem, 1 = almost never, 2 = sometimes, 3 = often and 4 = almost always). Items are linearly transformed to a 0-100 scale, so that higher scores indicate better quality of life.
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 20
units on a scale | 1.0 [-4.6 to 6.6]

30. Secondary Outcome: Changes in Physical Quality of Life From Baseline to 3 Months
Description: To examine the effects of waitlist intervention on quality of life, physical domain, at baseline and 3 months using Pediatric Quality of Life Inventory (PedsQL; UK version 4). The self-report scale had a five-point response scale (0 = never a problem, 1 = almost never, 2 = sometimes, 3 = often and 4 = almost always). Items are linearly transformed to a 0-100 scale, so that higher scores indicate better quality of life.
Time Frame: Baseline and 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 21
units on a scale | 4.0 [-1.7 to 9.8]

31. Secondary Outcome: Changes in Emotional Quality of Life From Baseline to 6 Months
Description: To examine the effects of waitlist intervention on quality of life, emotional domain, at baseline and 6 months using Pediatric Quality of Life Inventory (PedsQL; UK version 4). The self-report scale had a five-point response scale (0 = never a problem, 1 = almost never, 2 = sometimes, 3 = often and 4 = almost always). Items are linearly transformed to a 0-100 scale, so that higher scores indicate better quality of life.
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 20
units on a scale | 9.7 [-0.2 to 19.7]

32. Secondary Outcome: Changes in Emotional Quality of Life From Baseline to 3 Months
Description: To examine the effects of waitlist intervention on quality of life, emotional domain, at baseline and 3 months using Pediatric Quality of Life Inventory (PedsQL; UK version 4). The self-report scale had a five-point response scale (0 = never a problem, 1 = almost never, 2 = sometimes, 3 = often and 4 = almost always). Items are linearly transformed to a 0-100 scale, so that higher scores indicate better quality of life.
Time Frame: Baseline and 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 21
units on a scale | 6.5 [-3.4 to 16.3]

33. Secondary Outcome: Changes in School Quality of Life From Baseline to 6 Months
Description: To examine the effects of waitlist intervention on quality of life, school domain, at baseline and 6 months using Pediatric Quality of Life Inventory (PedsQL; UK version 4). The self-report scale had a five-point response scale (0 = never a problem, 1 = almost never, 2 = sometimes, 3 = often and 4 = almost always). Items are linearly transformed to a 0-100 scale, so that higher scores indicate better quality of life.
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 20
units on a scale | 6.9 [0.2 to 13.7]

34. Secondary Outcome: Changes in School Quality of Life From Baseline to 3 Months
Description: To examine the effects of waitlist intervention on quality of life, school domain, at baseline and 3 months using Pediatric Quality of Life Inventory (PedsQL; UK version 4). The self-report scale had a five-point response scale (0 = never a problem, 1 = almost never, 2 = sometimes, 3 = often and 4 = almost always). Items are linearly transformed to a 0-100 scale, so that higher scores indicate better quality of life.
Time Frame: Baseline and 3 Months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 21
units on a scale | 8.3 [0.6 to 16.1]

35. Secondary Outcome: Changes in Psychosocial Quality of Life From Baseline to 6 Months
Description: To examine the effects of waitlist intervention on quality of life, psychosocial domain, at baseline and 6 months using Pediatric Quality of Life Inventory (PedsQL; UK version 4). The self-report scale had a five-point response scale (0 = never a problem, 1 = almost never, 2 = sometimes, 3 = often and 4 = almost always). Items are linearly transformed to a 0-100 scale, so that higher scores indicate better quality of life.
Time Frame: Baseline and 6 Months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 20
units on a scale | 6.5 [0.2 to 12.7]

36. Secondary Outcome: Changes in Psychosocial Quality of Life From Baseline to 3 Months
Description: To examine the effects of waitlist intervention on quality of life, psychosocial domain, at baseline and 3 months using Pediatric Quality of Life Inventory (PedsQL; UK version 4). The self-report scale had a five-point response scale (0 = never a problem, 1 = almost never, 2 = sometimes, 3 = often and 4 = almost always). Items are linearly transformed to a 0-100 scale, so that higher scores indicate better quality of life.
Time Frame: Baseline and 3 Months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 21
units on a scale | 6.3 [0.2 to 12.5]

37. Secondary Outcome: Insulin Resistance Index Changes
Description: Examine changes in insulin resistance index at baseline and 6 months. Insulin resistance index is calculated according to the formula: fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: insulin resistance index
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 11
insulin resistance index | -0.3 [-1.8 to 1.2]

38. Secondary Outcome: Changes in Fasting Blood Glucose From Baseline to 6 Months
Description: Examine changes in fasting blood glucose result changes at baseline and month 6 measured in nmol/L
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 13
mmol/L | -0.07 [-0.25 to 0.11]

39. Secondary Outcome: Changes in 120 Minute Glucose Result in Oral Glucose Tolerance Test Measurements
Description: Examine changes in 120 minute glucose result changes in oral glucose tolerance test at baseline and month 6 measured in nmol/L.
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 13
mmol/L | -0.48 [-1.2 to 0.22]

40. Secondary Outcome: Changes in Fasting Lipid Measurements, High Density Lipoprotein (HDL), From Baseline to 6 Months
Description: Examine changes in fasting lipids, high density lipoprotein cholesterol (HDL), at month 6 measured in mg/dL
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 13
mmol/L | 0.06 [-0.03 to 0.15]

41. Secondary Outcome: Changes in Fasting Lipid Measurements, Low Density Lipoprotein (LDL), From Baseline to 6 Months
Description: Examine changes in fasting lipids, low density lipoprotein cholesterol (LDL), at month 6 measured in mg/dL
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 13
mmol/L | 0.11 [-0.16 to 0.38]

42. Secondary Outcome: Changes in Fasting Lipid Measurements, Triglycerides (TG), From Baseline to 6 Months
Description: Examine changes in fasting lipids, Triglycerides (TG), at month 6 measured in mg/dL
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 13
mmol/L | 0.05 [-1.20 to 0.23]

43. Secondary Outcome: Changes in Alanine Transaminase From Baseline to 6 Months
Description: Changes in Alanine transaminase from Baseline to 6 months measured in U/L
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: U/L
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 8
U/L | 11.9 [-5.9 to 29.6]

44. Secondary Outcome: Changes in Aspartate Transaminase From Baseline to 6 Months
Description: Changes in Aspartate transaminase from Baseline to 6 months, measured in U/L
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: U/L
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 8
U/L | 4.0 [-3.2 to 11.2]

45. Secondary Outcome: Changes in Disordered Eating on Dietary Restraint From Baseline to 6 Months
Description: To examine the effects of waitlist intervention on disordered eating at baseline and 6 months. Psychological dimensions of eating behaviors were determined using a validated self-reporting Eating Pattern Inventory for Children (EPI-C). The 20-item questionnaire assessed four dimensions ((dietary restraint, external eating, parental pressure to eat, and emotional eating). Responses to each item were listed on a 4-point Likert scale (1 = not at all, 2 = sometimes, 3 = mostly, 4 = always). Higher scores are indicative of greater dietary restraint.
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: score on epi
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 20
score on epi | 0.00 [-0.23 to 0.23]

46. Secondary Outcome: Changes in Disordered Eating, Dietary Restraint From Baseline to 3 Months
Description: To examine the effects of waitlist intervention on disordered eating at baseline and 3 months. Psychological dimensions of eating behaviors were determined using a validated self-reporting Eating Pattern Inventory for Children (EPI-C). The 20-item questionnaire assessed four dimensions ((dietary restraint, external eating, parental pressure to eat, and emotional eating). Responses to each item were listed on a 4-point Likert scale (1 = not at all, 2 = sometimes, 3 = mostly, 4 = always). Higher scores are indicative of greater dietary restraint.
Time Frame: Baseline and 3 months
Measure: Mean (95% Confidence Interval); unit: score on EPI
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 21
score on EPI | 0.033 [-0.15 to 0.21]

47. Secondary Outcome: Changes in Disordered Eating, External Eating From Baseline to 6 Months
Description: To examine the effects of waitlist intervention on External Eating dimension on disordered eating at baseline and 6 months. Psychological dimensions of eating behaviors were determined using a validated self-reporting Eating Pattern Inventory for Children (EPI-C). The 20-item questionnaire assessed four dimensions ((dietary restraint, external eating, parental pressure to eat, and emotional eating). Responses to each item were listed on a 4-point Likert scale (1 = not at all, 2 = sometimes, 3 = mostly, 4 = always). Higher scores are indicative of greater dietary restraint.
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: score on EPI
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 20
score on EPI | -0.19 [-0.50 to 0.12]

48. Secondary Outcome: Changes in Disordered Eating, External Eating From Baseline to 3 Months
Description: To examine the effects of waitlist intervention on External Eating dimension on disordered eating at baseline and 3 months. Psychological dimensions of eating behaviors were determined using a validated self-reporting Eating Pattern Inventory for Children (EPI-C). The 20-item questionnaire assessed four dimensions ((dietary restraint, external eating, parental pressure to eat, and emotional eating). Responses to each item were listed on a 4-point Likert scale (1 = not at all, 2 = sometimes, 3 = mostly, 4 = always). Higher scores are indicative of greater dietary restraint.
Time Frame: Baseline and 3 months
Measure: Mean (95% Confidence Interval); unit: score on EPI
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 21
score on EPI | -0.087 [-0.44 to 0.27]

49. Secondary Outcome: Changes in Disordered Eating, Parental Pressure to Eat, From Baseline to 6 Months
Description: To examine the effects of waitlist intervention on Parental Pressure to Eat dimension on disordered eating at baseline and 6 months. Psychological dimensions of eating behaviors were determined using a validated self-reporting Eating Pattern Inventory for Children (EPI-C). The 20-item questionnaire assessed four dimensions ((dietary restraint, external eating, parental pressure to eat, and emotional eating). Responses to each item were listed on a 4-point Likert scale (1 = not at all, 2 = sometimes, 3 = mostly, 4 = always). Higher scores are indicative of greater dietary restraint.
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: score on EPI
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 20
score on EPI | 0.018 [-0.30 to 0.33]

50. Secondary Outcome: Changes in Disordered Eating, Parental Pressure to Eat, From Baseline to 3 Months
Description: To examine the effects of waitlist intervention on Parental Pressure to Eat dimension on disordered eating at baseline and 3 months. Psychological dimensions of eating behaviors were determined using a validated self-reporting Eating Pattern Inventory for Children (EPI-C). The 20-item questionnaire assessed four dimensions ((dietary restraint, external eating, parental pressure to eat, and emotional eating). Responses to each item were listed on a 4-point Likert scale (1 = not at all, 2 = sometimes, 3 = mostly, 4 = always). Higher scores are indicative of greater dietary restraint.
Time Frame: Baseline and 3 months
Measure: Mean (95% Confidence Interval); unit: score on EPI
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 21
score on EPI | 0.116 [-0.12 to 0.35]

51. Secondary Outcome: Changes in Disordered Eating, Emotional Eating, From Baseline to 6 Months
Description: To examine the effects of waitlist intervention on Emotional Eating dimension on disordered eating at baseline and 6 months. Psychological dimensions of eating behaviors were determined using a validated self-reporting Eating Pattern Inventory for Children (EPI-C). The 20-item questionnaire assessed four dimensions ((dietary restraint, external eating, parental pressure to eat, and emotional eating). Responses to each item were listed on a 4-point Likert scale (1 = not at all, 2 = sometimes, 3 = mostly, 4 = always). Higher scores are indicative of greater dietary restraint.
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: score on EPI
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 20
score on EPI | 0.171 [-0.15 to 0.49]

52. Secondary Outcome: Changes in Disordered Eating, Emotional Eating, From Baseline to 3 Months
Description: To examine the effects of waitlist intervention on Emotional Eating dimension on disordered eating at baseline and 3 months. Psychological dimensions of eating behaviors were determined using a validated self-reporting Eating Pattern Inventory for Children (EPI-C). The 20-item questionnaire assessed four dimensions ((dietary restraint, external eating, parental pressure to eat, and emotional eating). Responses to each item were listed on a 4-point Likert scale (1 = not at all, 2 = sometimes, 3 = mostly, 4 = always). Higher scores are indicative of greater dietary restraint.
Time Frame: Baseline and 3 months
Measure: Mean (95% Confidence Interval); unit: score on EPI
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 21
score on EPI | 0.00 [-0.34 to 0.34]

53. Secondary Outcome: Metabolomic Profile Changes From Baseline to 6 Months (BCAA)
Description: Examine changes in branched chain amino acid(BCAA) at baseline and month 6. Metabolites to be analysed include BCAA which is a combination of isoleucine, leucine, valine. All metabolites concentrations will be reported in micro mol per litre
Time Frame: baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: micro mol/L
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 13
micro mol/L | 15.06 [-54.95 to 85.07]

54. Secondary Outcome: Metabolomic Profile Changes From Baseline to 6 Months (AAA)
Description: Examine changes in aromatic amino acid (AAA) at baseline and month 6. Metabolites to be analysed include AAA which is a combination of phenylalanine and tyrosine. All metabolites concentrations will be reported in micro mol per litre.
Time Frame: baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: micro mol/L
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 13
micro mol/L | 1.70 [-22.11 to 25.50]

ADVERSE EVENTS:
Time Frame: 6 months
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed. No Self reported adverse event.
Arm/Group | Mobile Health Application
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: Informed Consent Form (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT03561597/Prot_SAP_ICF_000.pdf
  • Informed Consent Form: Informed Consent Form (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT03561597/ICF_001.pdf